CLINICAL TRIAL: NCT07060768
Title: The Effect of Mandala Coloring on Perinatal Grief and Psychological Resilience Levels in Women Experiencing Perinatal Loss: A Randomized Controlled Trial
Brief Title: The Effect of Mandala Coloring on Perinatal Grief and Psychological Resilience Levels in Women Experiencing Perinatal Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Elif Balkan, Research Assistant, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EBYalova
Record Dates: First submitted 2025-06-21; First posted 2025-07-11 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Perinatal Loss
Keywords: perinatal loss; resilience; perinatal grief

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will have mandala coloring intervention
  Interventions: Other: Mandala Coloring
- Control (No Intervention): This arm will not receive any intervention

INTERVENTIONS:
Other: Mandala Coloring — Mandala coloring at least 20 minutes each day. Totally 10 days intervention
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to evaluate if mandala colouring helps to decrease grief symptoms and increase resilience in women who experienced perinatal loss.

The main questions are:

Does mandala coloring decrease perinatal grief symptoms? Does mandala coloring increase resilience?

Researchers will compare mandala coloring intervention with standard perinatal loss nursing care to evaluate if mandala coloring works to decrease grief symptoms.

Participants will:

Answer some questionnaires and scales, and do mandala coloring at least for 20 minutes for 10 days after perinatal loss experience.

ELIGIBILITY:
Inclusion Criteria:

* Experienced perinatal loss (neonatal death, fetal death, abortion) within the last six weeks

Exclusion Criteria:

* Serious psychological problem that requires intervention with the recommendation of a psychiatrist, such as having a previous mental disorder or use of antidepressants.
* Practicing alternative methods such as yoga, meditation, acupuncture

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender people identify with the gender that aligns with the sex they were assigned at birth
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Perinatal Grief | 1st day to 10th day
  Perinatal Grief will be assessed via Perinatal Grief Scale. The scale is a 5-point Likert-type scale and responses range from "strongly agree to strongly disagree". The scale includes three sub-dimensions: "active grief", "difficulty coping" and "hopelessness". The total number of items in the scale is 32. Items 11 and 32 of the scale have a positive sentence structure. These items are answered in reverse. While the total grief score that can be obtained from the scale varies between 32-160, the scores that can be obtained for each sub-dimension seperately.
  As the total perinatal grief score and the total score obtained from the sub-dimensions increase, it is determined that the individual's grief level is higher.
Perinatal Grief Intensity | 1st day to 10th day
  Will be assessed via Perinatal Grief Intensity Scale. The scale consists of 14 items, rated on a 4-point Likert-type scale from strongly agree to strongly disagree, and three sub-dimensions: "reality", "confrontation with others", and "adaptation". The scale contains both positive and negative expressions. Therefore, items 1, 2, 3, and 6 are evaluated as reverse items in the scoring of the scale. When calculating the scores of the sub-dimensions, the score obtained from each item is added up and divided by the number of items in the sub-dimension. Thus, a total score between 1 and 4 is obtained from each sub-dimension. The following formula is used for the total score:
  3.08 + (0.41 x reality sub-dimension mean score) - (0.2 x confrontation sub-dimension mean score) - (0.15 x harmony sub-dimension mean score) The score that can be obtained from the scale varies between 2.09 - 4.37. It is predicted that the intensity of grief that will be experienced increases as the score increases

SECONDARY OUTCOMES:
Resilience | 1st day and 10th day
  Will be assessed via Resilience Scale for Adults. The scale has a schematic evaluation with five boxes. The scale consists of six factors titled 'Self-perception, 'Future perception,' 'Structural style,' 'Social competence,' 'Family harmony,' and 'Social resources,' and contains a total of 33 items. Cronbach's alpha coefficient of the sub-dimensions of the scale varies between 0.75-0.86

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared publicly due to ethical restrictions. But authors may share IPD with researchers who reach out to the authors for data sharing with necessary reasons

REFERENCES:
- [Background] Hutti MH, dePacheco M, Smith M. A study of miscarriage: development and validation of the Perinatal Grief Intensity Scale. J Obstet Gynecol Neonatal Nurs. 1998 Sep-Oct;27(5):547-55. doi: 10.1111/j.1552-6909.1998.tb02621.x. PMID 9773366
- [Background] Kones MO, Kaydırak MM, Aslan E, Yildiz H. The Perinatal Grief Scale (33-item short version): validity and reliability of the Turkish version. Anadolu Psikiyatri Derg. 2017; 18(3): 231-236. doi:10.5455/apd.234509.
- [Background] Toedter LJ, Lasker JN, Alhadeff JM. The Perinatal Grief Scale: development and initial validation. Am J Orthopsychiatry. 1988 Jul;58(3):435-49. doi: 10.1111/j.1939-0025.1988.tb01604.x. PMID 3407734